CLINICAL TRIAL: NCT00947232
Title: The Effectiveness of Physical Activity for Major Depression in People Aging With Multiple Sclerosis or Spinal Cord Injury
Brief Title: Motivational Interviewing to Increase Physical Activity to Treat Depression in People Aging With MS or SCI
Acronym: inMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Charles Bombardier, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36020-J; H133B080024
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis; Spinal Cord Injury
Keywords: major depressive disorder; physical activity; aging with physical disability; motivational interviewing
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries; Depressive Disorder, Major; Motor Activity | interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing (Experimental): Motivational interviewing for people aging with multiple sclerosis or spinal cord injury to increase physical activity and decrease depression.
  Interventions: Behavioral: Motivational interviewing
- Education (Active Comparator): Education about physical activity for people aging with multiple sclerosis or spinal cord injury to decrease depression.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing, a proven counseling method that centers on individual goals and motivations, to increase exercise and decrease depression.
  Arms: Motivational interviewing
Behavioral: Education — Educational intervention about the benefits of physical activity to decrease depression for people aging with multiple sclerosis or spinal cord injury.
  Arms: Education

SUMMARY:
This study compares two approaches to helping people who are aging with MS or SCI and are experiencing depressed mood to become more physically active. The study is carried out entirely by telephone. There is no need to travel and participants may reside anywhere within the United States. We will examine the effects of the intervention on overall physical activity, mood, pain, fatigue and general health. Participants will complete surveys over the phone throughout the study and wear an activity monitor 3 times. The study is 6 months in length and participants may receive up to $120 for their time and effort.

DETAILED DESCRIPTION:
People aging with disabilities such as spinal cord injury (SCI) or multiple sclerosis (MS) report high rates of major depression. Depression frequently adds to the disabilities and suffering in these populations. Few definitive studies of depression treatments have been done in people with MS and none in SCI. There are several reasons to explore novel treatments for major depression in these groups. First, standard treatments, such as antidepressant medications, may not be as effective in people with neurological disabilities. Next, people with physical disabilities tend to be inactive. Lack of physical activity has been positively correlated with higher levels of depression. Longitudinal data and treatment trials suggest that increased physical activity is related to improved mood. Controlled trials show that increased exercise and physical activity can be effective treatments for major depression in nondisabled older adults. Previous research by the investigators' group suggests that people with MS are quite interested in exercise and that exercise is a safe and effective treatment for depression in younger, less disabled people with MS. Exercise may have widespread benefits for people with MS or SCI. Finally, exercise or increased physical activity represents a low cost, non-stigmatizing, highly accessible potential treatment for depression in people with physical disabilities. In this study the investigators will determine whether a relatively brief telephone-based intervention to promote physical activity is an effective treatment for major depression in people aging with MS or SCI. The investigators define "aging" as chronological age greater than 45 years old.

ELIGIBILITY:
Inclusion Criteria:

* aged at least 45 years old
* self-report diagnosis of MS or SCI
* meeting SCID requirements for Major Depressive Disorder (MDD) or dysthymia
* MS: EDSS between 4.0 and 8.0
* SCI: ASIA A-D injury level at or below C4 and they have upper extremity function sufficient to propel a manual wheelchair
* meeting PHQ-9 measure cut-off for depression by scoring more than 10 on the measure
* currently inactive (exercising less than 150 minutes per week)
* response form received from participants' doctor declaring exercise safe for the subject.

Exclusion Criteria:

* significant cognitive impairment
* pressure ulcers on sitting surfaces (or another condition that precludes sitting
* significant obesity (>160% of ideal body weight)
* significant risk factors for beginning moderate physical activity measured with the PAR-Q
* response form received from participants' doctor declaring exercise unsafe for the subject
* a self-reported history of significant Uthoff's effect for those with MS
* psychiatric contraindications such as bipolar disorder, psychosis, active suicidal ideation with intent or plan, or current alcohol or drug dependence. We will include people who remain depressed but are on stable doses of antidepressant medications.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
HAM-D | Baseline, weeks 4, 6, 8, 12, and 24
  17-item interview based depression severity measure

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline, weeks 4, 6, 8, 12, and 24
  self-reported measure of weekly light, moderate and vigorous physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bombardier, PhD, Principal Investigator — University of Washington; Mark Jensen, PhD, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website for the Aging Rehabilitation Research and Training Center — http://agerrtc.washington.edu